CLINICAL TRIAL: NCT02021149
Title: Enhancing Psychotherapy for Mood Disorders With Whole Body Hyperthermia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator transferred to the University of Wisconsin - Madison
Sponsor: Charles (Chuck) Raison (Other)
Responsible Party: Sponsor-Investigator, Charles (Chuck) Raison, Associate Professor, Department of Psychiatry (College of Medicine) and the Norton School of Family and Consumer Sciences, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-0614
Record Dates: First submitted 2013-11-26; First posted 2013-12-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Whole Body Hyperthermia; Psychotherapy; Therapist and patient alliance
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Psychotherapy; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Psychotherapy and Questionnaire Group (Other): Participants in this arm will have their regular psychotherapy sessions with their psychotherapist and will, prior to each session, fill out study related questionnaires.
  Interventions: Behavioral: Psychotherapy; Other: Questionnaires
- High intensity whole-body infrared heating and Psychotherapy. (Experimental): Subjects will have weekly psychotherapy sessions and fill out study questionnaires. The participant's 4th psychotherapy session will be conducted while the patient undergoes the WBH intervention where subjects will be induced to levels of heat that increases core body temperature to approximately 37.5-38.5 °C.temperature.
  Interventions: Device: High intensity whole-body infrared heating; Behavioral: Psychotherapy; Other: Questionnaires
- Low intensity whole-body infrared heating and Psychotherapy (Sham Comparator): Subjects will have weekly psychotherapy sessions and fill out study questionnaires. The participant's 4th psychotherapy session will be conducted while the patient undergoes WBH-control where subjects will be induced to levels of heat that causes only a minor increase in body temperature.
  Interventions: Behavioral: Psychotherapy; Other: Questionnaires; Device: Low intensity whole-body infrared heating

INTERVENTIONS:
Device: High intensity whole-body infrared heating — The Whole Body Hyperthermia system uses water-filtered infrared-A (wIRA) heat radiation. The rise in the body's core temperature is correspondingly rapid and well-tolerated. There are two phases of the thermal challenge, 1) Irradiation phase during which the patient lies recumbent with his/her head positioned outside the tent. The wIRA irradiators are arranged above the exposed upper part of the body; and 2) Heat retention phase during which the patient lies in the chamber with the walls of the tent positioned to retain heat. Core body temperatures will be raised to those comparable to a mild fever 37.8-38.5°C.
  Arms: High intensity whole-body infrared heating and Psychotherapy.
Behavioral: Psychotherapy — Weekly psychotherapy using cognitive behavioral therapy sessions with a therapist.
Other: Questionnaires — Weekly questionnaires to assess changes in mood, perceptions of self and perceptions of effectiveness of the therapist/patient bond will be administered.
Device: Low intensity whole-body infrared heating — Attenuated heating using only heating coils at the bottom of the Heckel device. This results in only a minor increase in skin temperature and no increase in core body temperature. The participant will still feel heat and will see similar lighting and hear similar sounds as those occurring during actual WBH, and will be in the chamber for the same period of time.
  Arms: Low intensity whole-body infrared heating and Psychotherapy

SUMMARY:
According to the 2005 National Comorbidity Survey-Replication study, approximately 20.9 million American adults, or 9.5 percent of the population over the age of 18 suffer from mood disorders including major depressive disorder, chronic, mild depression and bipolar disorder. Major depressive disorder (MDD) is predicted to be the second leading cause of disability worldwide by the year 2020; sub-clinical mood disturbances impact many additional people and are a major reason people seek psychotherapy services. The economic burden of depression in the United States is significant: $83.1 billion in 2000 and increasing. Much of this burden comes from the high rate of sub-optimal treatment outcomes associated with the disorder. Indeed, only 50% of MDD patients recover in less than 12 weeks with adequate treatment, and up to 20% of patients will fail to adequately respond to all currently available interventions. Moreover, current treatments come at the cost of significant central nervous system (CNS) side effects, further highlighting the need for more effective treatments with fewer side effects. To address these pressing clinical issues, the investigators will conduct a placebo controlled, clinical trial to determine if Whole Body Hyperthermia (WBH) enhances the effects of psychotherapy compared to psychotherapy alone in medically healthy patients with moderate to severe mood disorders. The investigators plan to recruit a sample of 24 medically healthy individuals with mood problems who will be randomized to examine whether WBH enhances the effects of psychotherapy. To determine acute and sustained effects of WBH +psychotherapy on mood disorders, the study will include basic psychiatric questionnaire-based assessments at three therapy sessions prior to a single session conducted while receiving one of two intensities of WBH treatment. Subjects who elect not to conduct a therapy session in the WBH chamber will still be able to complete study questionnaires at all therapy sessions. This study challenges the existing paradigm by determining if peripheral afferent sensory pathways can be accessed to enhance the treatment of mood disorders and thus avoid problems of exposing all of the brain to non-selective drugs.

DETAILED DESCRIPTION:
Our research group has observed in an open trial that a single session of whole body hyperthermia (WBH) induced rapid antidepressant effects that persisted for at least a week in patients with major depression (MDD) severe enough to warrant inpatient hospitalization. In addition to reducing depression, the single session of WBH induced a prolonged reduction in mean core body temperature, consistent with basic science data from our group suggesting that hyperthermia activates a skin-to-brain pathway that targets specific serotonergic nuclei in the raphe. In animal models, these nuclei have been shown to be important for mood and body temperature regulation. Consistent with this known anatomy in our preliminary study in depressed patients, reductions in core body temperature were highly correlated with reductions in depressive symptoms over the same time period (one week post WBH). Moreover, patients with higher mean core body temperature prior to treatment had enhanced antidepressant effects. Because increased body temperature is an outcome of poor functioning in the skin-to-brain pathway activated by WBH our data suggests that WBH may actually sensitize this pathway in ways that promote changes in brain functioning known to promote emotional well-being. The results of our first open trial have encouraged us to conduct a larger, more rigorous placebo-controlled, double blind study of WBH for MDD, which is currently underway at the University of Arizona Medical School.

In addition to impacting depressive symptoms and body temperature, The investigators have observed that WBH induces striking increases in prosocial and self-disclosing behavior in many individuals. This effect initiates in the heating phase of the treatment and culminates at maximum body temperature. Importantly, our observations thus far suggest that this prosociality only occurs when the person in the hyperthermia box is accompanied by someone he/she knows to at least some degree. For example, a recent subject was silent during his initial WBH treatment in which he was attended by one of our staff that he had never met. He elected to get a repeat WBH session. The same "attendant" was present for this second WBH session, and during this session the patient became strikingly talkative and without prompting self-disclosed a range of very intimate personal issues related to his depression, such as a previously undisclosed history of childhood sexual abuse.

The goal of the current proposal is to conduct a pilot study to evaluate whether this observed prosocial effect of WBH might be employed to accelerate and deepen the formation of therapeutic alliance in patients undergoing an 8-12 session course of cognitive behavioral psychotherapy (CBT). Our study design will also more rigorously test our clinical observation about the prosocial effects of WBH. In addition to potentially enhancing psychotherapeutic outcomes, the current study may provide data relevant to larger issues related to the near universal use of hyperthermia in indigenous cultures around the world for spiritual and health purposes.

ELIGIBILITY:
Inclusion Criteria for Psychotherapy and Questionnaire Group:

- The only inclusion criteria for this group is that they are deemed eligible to receive psychotherapy at the Psychology Department Clinic, are fluent in English and are interested in participating in the study. There are no specific exclusion criteria for this study group.

Inclusion Criteria for WBH Psychotherapy Group:

* Male or female outpatients aged 18-65.
* Able to understand the nature of the study and able to provide written informed consent prior to conduct of any study procedures.
* Able to communicate in English with study personnel.
* For women of child-bearing potential (i.e., one who is biologically capable of becoming pregnant), must be willing to use a medically acceptable form of birth control or practice abstinence for the duration of her participation in the trial.

Exclusion Criteria:

* Any of the following diagnoses, as identified by the intake evaluation conducted or study assessments:
* A diagnosis claustrophobia severe enough that it would impair ability to be in the Heckel HT3000 hyperthermia device
* A current (or within 12 months prior to the Screening visit) diagnosis of Anorexia Nervosa or Bulimia Nervosa
* Subject has a medical condition or disorder that:
* Is unstable and clinically significant, or:
* Could interfere with the accurate assessment of safety or efficacy of treatment, including:
* individuals who are using prescription drugs that may impair thermoregulatory cooling, including diuretics, barbiturates, and beta-blockers, or antihistamines,
* individuals with cardiovascular conditions or problems (uncontrolled hypertension, congestive heart failure, or documented evidence of coronary artery disease)
* individuals with chronic conditions/diseases associated with a reduced ability initiate thermoregulatory cooling, including Parkinson's, multiple sclerosis, central nervous system tumors, and diabetes with neuropathy,
* hemophiliacs/individuals prone to bleeding,
* individuals with a fever the day of study intervention,
* individuals with hypersensitivity to heat,
* individuals with recent acute joint injury,
* individuals with enclosed infections, be they dental, in joints, or in any other tissues,
* Clinically significant, in the investigator's opinion, abnormal findings on screening laboratory tests or physical exam as presented to the research team.
* Use of any psychotropic medications for 2 weeks (8 weeks for fluoxetine) prior to initiation of the study, with the exception of hypnotic medications (zolpidem, zaleplon, eszopiclone).
* Need for any non-protocol psychotropic medication during the trial, with the exception of hypnotics used up to four nights per week.
* Women who are pregnant (HCG pregnancy test at screening, or lactating, or who plan to become pregnant during the study.
* Current participation in any clinical trial that might impact results of this one, which includes participation in another clinical trial for depression, as well as drug trials with agents that might affect mood or regulation of body temperature.
* Reasonable likelihood for non-compliance with the protocol for any other reason, in the opinion of the Investigator, prohibits enrollment of subject into the study.
* Obesity and overall size of subject. It will be up to the PI's discretion will consider BMI, waist circumference, and body fat composition when determining eligibility and safety of the individual.
* History of peripheral circulatory disease, for example peripheral vascular disease, deep vein thrombosis (DVT), or lymphedema.
* History of a cerebral vascular accident
* History of stroke, epilepsy or cerebral aneurisms
* Cancer in the last five years.
* Diabetes mellitus types I or II
* Any clinically significant autoimmune disease (compensated hypothyroidism allowed)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Change in depression scores over time [Inventory of Depressive Symptomatology-Self Report (IDS-SR)] | Intake Session and at therapy sessions every week thereafter (Weeks 2-12), including the session that occurs during the WBH/WBH-control intervention.
  Percentage change in scores between baseline and subsequent assessments will be assessed.
Change in Therapeutic bond / alliance | Intake Session and at therapy sessions every week thereafter (Weeks 2-12).
  Percentage change over time in the therapeutic alliance between patients and their therapists.

SECONDARY OUTCOMES:
Change in depression scores over time (OQ-45 Measurement) | Intake Session and at therapy sessions every week thereafter (Weeks 2-12), including the session that occurs during the WBH/WBH-control intervention.
  Percent change in scores between baseline and subsequent assessments will be assessed.
Change in Vitality | Intake Session and at therapy sessions every week thereafter (Weeks 2-12), including the session that occurs during the WBH/WBH-control intervention.
  Percent change in scores between baseline and subsequent assessments will be assessed using a vitality scale.
Change in Positive and Negative Affect | Intake Session and at therapy sessions every week thereafter (Weeks 2-12), including the session that occurs during the WBH/WBH-control intervention.
  Percent change in positive and negative affect will be assessed between baseline and subsequent assessments using the Positive and Negative Affect Schedule (PANAS)
Change in relationship with psychotherapist | Intake Session and at therapy sessions every week thereafter (Weeks 2-12), including the session that occurs during the WBH/WBH-control intervention.
  The investigators will use qualitative coding of psychotherapy sessions recorded at each psychotherapy session to assess whether WBH + psychotherapy affects and strengthens the ways in which patients relate to their psychotherapist and determined whether or not it enhances psychotherapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — University of Arizona, Department of Psychiatry, College of Medicine; David Sbarra, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States